CLINICAL TRIAL: NCT05409989
Title: MicroVention, Inc. Flow Re-Direction Endoluminal Device X (FRED™ X™) Post-Approval Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL11023
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Flow Re-Direction Endoluminal Device X (Other): FRED™ X™ device
  Interventions: Device: FRED™ X™

INTERVENTIONS:
Device: FRED™ X™ — The FRED™ X™ System is indicated for use in the internal carotid artery from the petrous segment to the terminus for the endovascular treatment.
  Other Names: Flow Re-Direction Endoluminal Device X

SUMMARY:
The objective of this study is to generate contemporaneous clinical data to facilitate a reasonable comparison of the performance of the FRED™ X™ device with the performance of the FRED™ device. The data generated from this study will be compared to the safety and effectiveness of the FRED™ device by meeting the same performance goals (PGs) established for the FRED™ pivotal study.

ELIGIBILITY:
Inclusion Criteria:

Subjects for this study must meet ALL the following criteria:

1. Subject has single target aneurysm in the internal carotid artery from petrous segment to the terminus of the internal carotid artery.
2. The parent artery diameter must be 2.0 - 5.0 mm distal and/or proximal to the target intracranial aneurysm.
3. Negative pregnancy test (serum or urine) in a female subject who has had menses in the last 18 months.
4. Subject commits to return to the investigational site for the 30- day, 6-month, 12-month, 2-year, 3-year, and 5-year follow-up evaluations.
5. The subject or his/her authorized representative must sign the IRB-approved written informed consent form prior to the start of any study procedures.
6. The subject has a modified Rankin Scale (mRS) ≤ 2.
7. The subject has a wide-necked ( ≥4mm or dome-to-neck ratio <2) saccular or fusiform aneurysm.

Exclusion Criteria:

Subjects shall be excluded from the study if ANY of the following conditions exist:

1. Subject who suffers from a subarachnoid hemorrhage in the last 60 days.
2. Subject who suffers from intracranial hemorrhage in the last 30 days.
3. Subject who presents with an intracranial mass or currently undergoing radiation therapy for carcinoma of the head or neck region.
4. Subject with symptomatic extracranial or intracranial stenosis of the parent artery (>50%) proximal to the target aneurysm.
5. Subject with an irreversible bleeding disorder, a platelet count < 100 x 103 cells/mm3 or known platelet dysfunction or a contraindication to or inability to tolerate anticoagulants/antiplatelet agents or thrombolytic drugs.
6. Subject with history of major bleeding disorder (based on coagulation profile and platelet count) and/or subject presents with signs of active bleeding.
7. Subject with known hypersensitivity to any component of the treatment device that cannot be medically controlled.
8. Subject with documented contrast allergy, or other condition that prohibits imaging.
9. Evidence of active bacterial infection at the time of treatment.
10. Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within 3 months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction less than 30%.
11. Subject with a pre-existing stent in place at the target aneurysm.
12. Subject who is unable to complete the required follow-ups.
13. Subject who is pregnant, breastfeeding, or of childbearing potential and unwilling to prevent pregnancy during their participation in the study.
14. Subject has a serious or life-threatening comorbidity that could confound study results and/or prevent completion of 5-year followup.
15. Subject is enrolled in another device or drug study in which participation could confound study results.
16. Subject has absent femoral pulses or other condition preventing femoral access, or is planned to be treated using a radial access approach.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint Part 1: Proportion of subjects that experience either Death or major stroke within 30 days post-procedure. | 30-days
  Major stroke is defined as a new neurological event that persists for >24 hours and results in a ≥4-point increase in the NIHSS score compared to baseline or compared to any subsequent lower score.
Primary Safety Endpoint Part 2: Proportion of subjects that experience neurological death or major ipsilateral stroke within 12 months post-procedure. | 12 months
  A major ipsilateral stroke is defined as that occurring within the vascular distribution of the stented artery. Neurological death is defined as a death which has been adjudicated by an independent clinical events committee to have directly resulted from a neurologic cause.
Primary Effectiveness Endpoint: The percent of subjects with (1) complete (100%) occlusion of the target aneurysm and ≤50% stenosis of the parent artery at the target IA, and (2) in whom an alternative treatment of the target IA had not been performed. | 12 months
  (1) Complete (100%) occlusion of the target aneurysm is assessed utilizing the Raymond-Roy Scale (Raymond Roy Class 1) and ≤50% stenosis of the parent artery at the target IA), and in whom an alternative treatment of the target IA had not been performed. The study will utilize independent Core Laboratory to adjudicate all angiographic outcomes, including aneurysm occlusion status and parent artery stenosis. (2) Alternative treatment is defined as re-treatment of the target aneurysm with an alternative treatment modality including open repair, endovascular placement of an additional stent or treatment of in-stent stenosis.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Memorial Healthcare Systems, Hollywood, Florida
  - Orlando Health, Orlando, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Baptist Healthcare System, Louisville, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - Ochsner Health, New Orleans, Louisiana
  - The Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Brigham Incorporated, Boston, Massachusetts
  - UMass Memorial Health, Worcester, Massachusetts
  - Albany Medical Center, Albany, New York
  - University at Buffalo, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - Mount Sinai, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas